CLINICAL TRIAL: NCT01316276
Title: Long Term Safety and Tolerability Study of Open-Label Liposomal Amikacin for Inhalation (ARIKACE™) in Cystic Fibrosis Patients With Chronic Infection Due to Pseudomonas Aeruginosa
Brief Title: Extension Study of Liposomal Amikacin for Inhalation in Cystic Fibrosis (CF) Patients With Chronic Pseudomonas Aeruginosa (Pa) Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR02-110
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Respiratory Infections; Pulmonary Cystic Fibrosis; cystic fibrosis transmembrane conductance regulator (CFTR); Anti-bacterial Agent; Arikayce; ALIS; LAI
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Infections | interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LAI (Experimental): 590 mg LAI QD via a PARI Investigational eFlow® Nebulizer System (eFlow®) for 28 days followed by a 28-day off-treatment period. This cycle (28 days on treatment, 28 days off treatment) was to be repeated for up to 12 cycles, divided into 2 periods of 6 cycles each (approximately 12 months each).
  Interventions: Drug: Liposomal amikacin for inhalation

INTERVENTIONS:
Drug: Liposomal amikacin for inhalation — * Liposomal amikacin for inhalation is provided as a sterile aqueous liposomal dispersion for inhalation via nebulization.
  * 590 mg of liposomal amikacin for inhalation is administered once daily using the PARI Investigational eFlow® Nebulizer.
  * Administration time is approximately 13 minutes.
  * Liposomal amikacin for inhalation will be administered in two consecutive extension periods, each consisting of 6 cycles for a total of 12 cycles. Each cycle consists of 28 days on-treatment followed by 28 days off-treatment.

SUMMARY:
The purpose of this study is to evaluate the long term safety and tolerability of Liposomal Amikacin for Inhalation (LAI) 590 mg once daily (QD) in Cystic Fibrosis patients with chronic infection due to pseudomonas aeruginosa. This long-term, open-label, multi-cycle extension study enrolled subjects who had successfully completed study TR02-108, were compliant with the study protocol, and did not meet any of the listed study discontinuation criteria. The safety and tolerability of LAI were evaluated for up to approximately 2 years.

DETAILED DESCRIPTION:
This was a long-term, open-label, multi-cycle extension study for patients in the Phase 3 study TR02-108 and TR02-109 who had successfully completed the 168-day study period and met study safety criteria. As this was a safety and tolerability long-term extension study, no sample size calculations were performed. All patients who completed TR02-108, were compliant with the study protocol, and did not meet any of the criteria listed for study discontinuation (safety reasons or non-compliance) were able to participate in this open-label study.

The end of study visit for TR02-108 was to serve as the baseline study visit (Day 1) for TR02-110 if the patient had signed the informed consent at least 4 days prior to the end of study visit and met all safety criteria for TR02-110. If the end of study visit was not used as the baseline visit, a separate baseline visit (Day 1) was to be performed within 14 days of completing TR02-108.

Patients were to receive a delivered dose of 590 mg LAI QD via a PARI Investigational eFlow® Nebulizer System (eFlow®) for 28 days followed by a 28-day off-treatment period. This cycle (28 days on treatment, 28 days off treatment) was to be repeated for up to 12 cycles. The study was implemented as 2 consecutive extension periods, each consisting of 48 weeks (approximately 12 months). Patients were re-consented for the second extension period at the completion of the first extension period. The total study period was up to 96 weeks (approximately 2 years).

During the first 28 days of treatment, patients were evaluated at the study site bi-weekly for safety, tolerability and efficacy. Thereafter, for the duration of the study, patients were evaluated at the study site on the first and last days of dosing during the on-treatment periods. During the study, starting with the off-treatment period of Cycle 1, patients were contacted by telephone once during every 28-day period to assess safety. A final site visit occurred 28 days after last dose of LAI. Arikace™, Arikayce™,Liposomal Amikacin for Inhalation (LAI), and Amikacin Liposome Inhalation Suspension (ALIS) may be used interchangeably throughout this study and other studies evaluating amikacin liposome inhalation suspension.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent or assent
* Subject has completed study TR02-108, and has been compliant with the study protocol
* Women of childbearing potential must agree to use reliable methods of contraception for the duration of the study

Key Exclusion Criteria:

* Subject met any of the listed criteria for study drug discontinuation in protocol TR02-108.
* Abnormal laboratory assessments including LFT (≥ 3× upper limit of normal [ULN]), serum creatinine (> 2× ULN) and absolute neutrophil count [ANC] (< 1000).
* Psychotic, addictive or other disorder limiting the ability to provide informed consent or to comply with study requirements.
* History of alcohol, medication or illicit drug abuse within the 6 months prior to consent.
* Smoking tobacco or any substance within 6 months prior to consent or anticipated inability to refrain from smoking throughout the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2012-10-05 (Actual); Primary Completion 2015-07-16 (Actual); Study Completion 2015-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Eagle, MD, Study Director — Insmed Incorporated
Locations (50):
- Vienna, Austria
- Belgium (4):
  - Antwerp
  - Brussels
  - Ghent
  - Leuven
- Bulgaria (4):
  - Pleven
  - Plovdiv
  - Sofia
  - Varna
- Canada (3):
  - Halifax
  - Hamilton
  - Vancouver
- Copenhagen, Denmark
- France (2):
  - Lille
  - Paris
- Germany (5):
  - Berlin
  - Essen
  - Hamburg
  - Hanover
  - München
- Greece (2):
  - Athens
  - Marousi
- Hungary (3):
  - Budapest
  - Debrecen
  - Szeged
- Dublin, Ireland
- Italy (5):
  - Brescia
  - Catania
  - Parma
  - Roma
  - Verona
- Utrecht, Netherlands
- Poland (7):
  - Gdansk
  - Lodz
  - Lublin
  - Poznan
  - Rabka-Zdrój
  - Rzeszów
  - Warsaw
- Belgrade, Serbia
- Slovakia (3):
  - Banská Bystrica
  - Bratislava
  - Košice
- Spain (3):
  - Barcelona
  - Madrid
  - Valencia
- United Kingdom (4):
  - Leeds
  - London
  - Nottingham
  - Penarth

REFERENCES:
- [Derived] Bilton D, Fajac I, Pressler T, Clancy JP, Sands D, Minic P, Cipolli M, Galeva I, Sole A, Quittner AL, Jumadilova Z, Ciesielska M, Konstan MW; CLEAR-110 Study Group. Long-term amikacin liposome inhalation suspension in cystic fibrosis patients with chronic P. aeruginosa infection. J Cyst Fibros. 2021 Nov;20(6):1010-1017. doi: 10.1016/j.jcf.2021.05.013. Epub 2021 Jun 16. PMID 34144923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study TR02-110 did not include any patients from Study TR02-109 since that study never enrolled patients.
Groups:
- LAI 590 mg QD: 590 mg LAI once a day (QD) via a PARI Investigational eFlow® Nebulizer System (eFlow®) for 28 days followed by a 28-day off-treatment period. This cycle (28 days on treatment, 28 days off treatment) was to be repeated for up to 12 cycles, divided into 2 periods of 6 cycles each (approximately 12 months each).
  Liposomal amikacin for inhalation (LAI): - Liposomal amikacin for inhalation is provided as a sterile aqueous liposomal dispersion for inhalation via nebulization.
  * 590 mg of liposomal amikacin for inhalation is administered once daily using the PARI Investigational eFlow® Nebulizer.
  * Administration time is approximately 13 minutes.
  * Liposomal amikacin for inhalation will be administered in two consecutive extension periods, each consisting of 6 cycles for a total of 12 cycles. Each cycle consists of 28 days on-treatment followed by 28 days off-treatment.
Period: Overall Study
Arm/Group | LAI 590 mg QD
Started | 206
Completed | 139
Not Completed | 67
Not completed — Death | 1
Not completed — Adverse Event | 19
Not completed — Withdrawal of consent | 24
Not completed — Lost to Follow-up | 1
Not completed — Other | 22

BASELINE CHARACTERISTICS:
Groups:
- LAI 590 mg QD: 590 mg LAI QD via a PARI Investigational eFlow® Nebulizer System (eFlow®) for 28 days followed by a 28-day off-treatment period. This cycle (28 days on treatment, 28 days off treatment) was to be repeated for up to 12 cycles, divided into 2 periods of 6 cycles each (approximately 12 months each).
  Liposomal amikacin for inhalation: - Liposomal amikacin for inhalation is provided as a sterile aqueous liposomal dispersion for inhalation via nebulization.
  * 590 mg of liposomal amikacin for inhalation is administered once daily using the PARI Investigational eFlow® Nebulizer.
  * Administration time is approximately 13 minutes.
  * Liposomal amikacin for inhalation will be administered in two consecutive extension periods, each consisting of 6 cycles for a total of 12 cycles. Each cycle consists of 28 days on-treatment followed by 28 days off-treatment.
Arm/Group | LAI 590 mg QD
Number analyzed (Participants) | 206
Age, Continuous [Mean (Standard Deviation); unit: years]
  Baseline age (years) | 21.0 (9.73)
Age, Customized [Count of Participants; unit: Participants]
  Age: Age group at baseline: 6 to 12 years | 37
  Age: Age group at baseline: >12 to 18 years | 62
  Age: Age group at baseline: >18 years | 107
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Caucasian (not of Hispanic origin) | 200
  Ethnicity: Hispanic | 5
  Ethnicity: African | 1
Geographic region [Count of Participants; unit: Participants]
  Western Europe / North America | 99
  Central Europe / Eastern Europe | 107

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Adverse Events (TEAEs) up to Day 672
Description: Treatment emergent adverse events including serious adverse events (SAE) and adverse events (AE) leading to permanent discontinuation of study drug
Time Frame: From Study Initiation up to Day 672
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | LAI 590 mg QD
Number analyzed (Participants) | 206
Participants
  Patients with ≥1 treatment-emergent AE | 183
  Patients with ≥ 1 serious AE | 92
  Patients with ≥1 AE leading to discontinuation | 21

2. Primary Outcome: Laboratory Abnormalities up to Day 672
Description: * Number of Subjects with Grade 3 or Higher Abnormalities in Clinical Laboratory Values
  * Number of Subjects with Grade 3 or Higher Hematology Laboratory Value Abnormalities
  * Number of Subjects with Grade 3 or Higher Chemistry Laboratory Value Abnormalities
Time Frame: Baseline, Day 377 and Day 672
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | LAI 590 mg QD
Number analyzed (Participants) | 206
Participants
  Baseline | 13
  Day 337/End of Study Year 1 | 8
  Day 672/End of Study Year 2 | 8
  Leukocytes (<2.0 × 109 /L) | 7
  Lymphocytes (<0.5 × 109 /L) | 12
  Neutrophils (<2.0 × 109 /L) | 23
  Platelets (<192 × 109 /L) | 1
  Alanine aminotransferase (>5.0 × ULN) | 2
  Aspartate aminotransferase (>5.0 × ULN) | 1
  Gamma-glutamyltransferase (>5.0 × ULN) | 2
  Indirect bilirubin (>3.0 × ULN) | 1
  Calcium (<2.1 mmol/L) | 1
  Serum glucose: >13.9 mmol/L | 14
  Serum glucose: < 2.2 mmol/L | 6
  Phosphate (<0.6 mmol/L) | 3
  Potassium: >6.0 mmol/L | 8
  Potassium: <3.6 mmol/L | 1
  Sodium: >155 mmol/L | 1
  Sodium: <130 mmol/L | 4
  Urate (> ULN with physiologic consequences) | 8

3. Primary Outcome: Acute Tolerability as Measured by Pulmonary Function Test (PFT) Changes Pre to Post Dose
Description: Number of Subjects with a >15% in Decline in Forced Expiratory Volume in 1 Second (FEV1) From Predose to Postdose
Time Frame: Day 1, Day 84, Day 196, Day 281, Day 337, Day 449, Day 532 and Day 644
Population: Safety Population
  Patients with missing values were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | LAI 590 mg QD
Number analyzed (Participants) | 206
Participants
  Day 1 | 6
  Day 84 | 6
  Day 196 | 1
  Day 281 | 5
  Day 337 | 5
  Day 449 | 6
  Day 532 | 2
  Day 644 | 3

4. Primary Outcome: Respiratory Rate: Change From Baseline to Day 672
Description: Respiratory rate was recorded at every visit as per standard practice at each investigational site.
Time Frame: From Study Initiation up to Day 672
Population: Safety Population Patients with missing data were excluded.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | LAI 590 mg QD
Number analyzed (Participants) | 133
breaths per minute | -0.8 (3.02)

5. Primary Outcome: Heart Rate: Change From Baseline From Day 672
Description: Pulse rate (after at least 5-minute rest) was recorded at every visit as per standard practice at each investigational site.
Time Frame: From Study Initiation up to Day 672
Population: Safety Population Patients with missing data were excluded.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | LAI 590 mg QD
Number analyzed (Participants) | 206
beats/min | -0.9 (12.46)

6. Primary Outcome: Systolic BP: Change From Baseline at Day 672
Description: Sitting blood pressure was recorded at every visit as per standard practice at each investigational site.
Time Frame: From Study Initiation up to Day 672
Population: Safety Population Patients with missing data were excluded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LAI 590 mg QD
Number analyzed (Participants) | 206
mmHg | 2.3 (11.39)

7. Primary Outcome: Diastolic BP: Change From Baseline at Day 672
Description: Sitting blood pressure was recorded at every visit as per standard practice at each investigational site.
Time Frame: From Study Initiation up to Day 672
Population: Safety Population Patients with missing data were excluded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LAI 590 mg QD
Number analyzed (Participants) | 206
mmHg | 1.5 (9.16)

8. Primary Outcome: Body Temperature: Change From Baseline at Day 672
Description: Body temperature was recorded at every visit as per standard practice at each investigational site.
Time Frame: From Study Initiation up to Day 672
Population: Safety Population Patients with missing data were excluded.
Measure: Mean (Standard Deviation); unit: Degrees Celcius
Arm/Group | LAI 590 mg QD
Number analyzed (Participants) | 206
Degrees Celcius | 0.03 (0.316)

9. Primary Outcome: Oxygen Saturation: Change From Baseline at Day 672
Description: Change in oxygen saturation as measured with pulse oximetry was performed via finger probes placed on the extremity opposite arterial lines and noninvasive blood pressure monitoring devices so that pulsatile flow was not interrupted.
Time Frame: From Study Initiation up to Day 672
Population: Safety Population Patients with missing data were excluded.
Measure: Mean (Standard Deviation); unit: Percent of Hemoglobin
Arm/Group | LAI 590 mg QD
Number analyzed (Participants) | 206
Percent of Hemoglobin | -0.1 (1.47)

10. Primary Outcome: Minimum Inhibitory Concentrations (MICs) for Pseudomonas Aeruginosa (Pa) and Burkholderia Species From Day 1 to Days 169, 337, 505 and 672
Description: Sputum was cultured for quantitative microbiological evaluation of Pa and Burkholderia species in designated regional central microbiology laboratories. A standard microbiology protocol was used for Pa culture and identification for each morphologically distinct Pa phenotype.
  Although planned in the Statistical Analysis Plan (SAP), MICs of amikacin Burkholderia species were not determined due to the small number of isolates with Burkholderia. In addition, susceptibility testing of isolates of Pa and Burkholderia species against a panel of commonly used antipseudomonal antibiotics was planned but was not performed.
  The results of the following analyses for Pa isolates are presented.
  * Frequency of MIC of Amikacin
  * Frequency of MIC of Tobramycin
  MIC50: lowest concentration of the antibiotic at which 50 % of the isolates were inhibited.
Time Frame: Day 1, Day 169, Day 337, Day 505 and Day 672
Population: Safety Population
  Patients with missing data were excluded.
Measure: Median (Full Range); unit: µg/mL
Arm/Group | LAI 590 mg QD
Number analyzed (Participants) | 206
µg/mL
  Amikacin MIC50: Day 1: number analyzed (Participants) | 180
  Amikacin MIC50: Day 1 | 16.000 [2.00 to 2048.00]
  Amikacin MIC50: Day 169: number analyzed (Participants) | 159
  Amikacin MIC50: Day 169 | 16.000 [1.00 to 2048.00]
  Amikacin MIC50: Day 337: number analyzed (Participants) | 143
  Amikacin MIC50: Day 337 | 16.000 [2.00 to 2048.00]
  Amikacin MIC50: Day 505: number analyzed (Participants) | 119
  Amikacin MIC50: Day 505 | 16.000 [0.25 to 2048.00]
  Amikacin MIC50: Day 672: number analyzed (Participants) | 109
  Amikacin MIC50: Day 672 | 16.000 [1.00 to 2048.00]
  Tobramycin MIC50: Day 1: number analyzed (Participants) | 180
  Tobramycin MIC50: Day 1 | 2.000 [0.25 to 1024.00]
  Tobramycin MIC50: Day 169: number analyzed (Participants) | 159
  Tobramycin MIC50: Day 169 | 2.000 [0.12 to 1024.00]
  Tobramycin MIC50: Day 337: number analyzed (Participants) | 143
  Tobramycin MIC50: Day 337 | 2.000 [0.25 to 1024.00]
  Tobramycin MIC50: Day 505: number analyzed (Participants) | 119
  Tobramycin MIC50: Day 505 | 2.000 [0.12 to 1024.00]
  Tobramycin MIC50: Day 672: number analyzed (Participants) | 109
  Tobramycin MIC50: Day 672 | 1.000 [0.12 to 1024.00]

11. Primary Outcome: Evaluation of Audiology
Description: Hearing was evaluated using air conduction [AC]. Bone conduction was required if the AC testing demonstrated a decrease of >20 decibels [dB]. Hearing loss was categorized using Common Terminology Criteria for Adverse Events as follows: GRADE 1 (best): Adults [A] on a Monitoring Program [MP]: Threshold shift of 15-25 dB; Pediatric [P]: Threshold shift >20 dB at 8 kilohertz (kHz). GRADE 2: [A] on a MP: Threshold shift of >25 dB; [A] not enrolled in MP: hearing loss; hearing aid/intervention not indicated; [P]: Threshold shift >20 dB at 4 kHz and above. GRADE 3: [A] enrolled in MP: Threshold shift of >25 dB; therapeutic intervention indicated; [A]: Not enrolled in MP: hearing aid/intervention; [P]: therapeutic intervention, including hearing aids: Threshold shift >20 dB at 3 kHz and above; additional speech-language related services. GRADE 4 (worst): [A]: Profound bilateral hearing loss; non-serviceable hearing; [P]: cochlear implant & additional speech-language related services.
Time Frame: Day 337 and Day 672
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | LAI 590 mg QD
Number analyzed (Participants) | 206
Participants
  Day 337/End of Study Day 337: None or minimal change | 133
  Day 337/End of Study Day 337: Grade 1 | 2
  Day 337/End of Study Day 337: Grade 2 | 0
  Day 337/End of Study Day 337: Grade 3 | 0
  Day 337/End of Study Day 337: Grade 4 | 0
  Day 337/End of Study Day 337: Indeterminate | 26
  Day 337/End of Study Day 337: Missing | 45
  Day 672/End of Study Day 672: None or minimal change | 120
  Day 672/End of Study Day 672: Grade 1 | 6
  Day 672/End of Study Day 672: Grade 2 | 0
  Day 672/End of Study Day 672: Grade 3 | 1
  Day 672/End of Study Day 672: Grade 4 | 0
  Day 672/End of Study Day 672: Indeterminate | 7
  Day 672/End of Study Day 672: Missing | 72

12. Primary Outcome: Change in Serum Creatinine Throughout the Study
Description: * Common Terminology Criteria for Adverse Events (CTCAE) Grade 1: > ULN-1.5 × ULN
  * CTCAE Grade 2: > 1.5 × ULN to 3.0 x ULN
Time Frame: Baseline, Day 337 and Day 672
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | LAI 590 mg QD
Number analyzed (Participants) | 206
Participants
  CTCAE Grade 1: Baseline: yes | 1
  CTCAE Grade 1: Baseline: no | 205
  CTCAE Grade 1: Day 337/End of Study Year 1: number analyzed (Participants) | 158
  CTCAE Grade 1: Day 337/End of Study Year 1: yes | 0
  CTCAE Grade 1: Day 337/End of Study Year 1: no | 158
  CTCAE Grade 1: Day 672/End of Study Year 2: number analyzed (Participants) | 131
  CTCAE Grade 1: Day 672/End of Study Year 2: yes | 0
  CTCAE Grade 1: Day 672/End of Study Year 2: no | 131
  CTCAE Grade 2: Baseline: yes | 0
  CTCAE Grade 2: Baseline: no | 206
  CTCAE Grade 2: Day 337/End of Study Year 1: number analyzed (Participants) | 158
  CTCAE Grade 2: Day 337/End of Study Year 1: yes | 0
  CTCAE Grade 2: Day 337/End of Study Year 1: no | 158
  CTCAE Grade 2: Day 672/End of Study Year 2: number analyzed (Participants) | 131
  CTCAE Grade 2: Day 672/End of Study Year 2: yes | 0
  CTCAE Grade 2: Day 672/End of Study Year 2: no | 131

13. Secondary Outcome: Percent Change in FEV1 Throughout the Study
Description: Percent Change From Baseline in Predose FEV1
Time Frame: Baseline, Day 337 and Day 672
Population: modified intention to treat (mITT) population
Measure: Mean (Standard Deviation); unit: Percent (%) change
Arm/Group | LAI 590 mg QD
Number analyzed (Participants) | 206
Percent (%) change
  Baseline | 2.104 (0.8650)
  Day 337: number analyzed (Participants) | 158
  Day 337 | 2.36 (14.359)
  Day 672: number analyzed (Participants) | 131
  Day 672 | 3.62 (18.485)

14. Secondary Outcome: Number of Subjects Experiencing a Protocol Defined Pulmonary Exacerbation
Description: For number of subjects to first protocol-defined pulmonary exacerbation, follow-up time began at the first dose of study drug (Day 1) and ended no later than Day 700 (28-day follow up).
Time Frame: From Study Initiation up to Day 700
Population: mITT
Measure: Number; unit: participants
Arm/Group | LAI 590 mg QD
Number analyzed (Participants) | 206
participants
  Number of patients with the event through Day 700 | 151
  Number censored | 55

15. Secondary Outcome: Number of Subjects Initiating Treatment.
Description: The number of subjects initiating antipseudomonal therapy for protocol-defined pulmonary exacerbation confirmed by the investigator, and for investigator-defined pulmonary exacerbation were summarized.
  The data presented below is the Frequency of Systemic or Inhaled Antipseudomonal Therapy for Protocol-defined Pulmonary Exacerbations Confirmed by Investigator
  - Time to First Use of Any New Antibiotic Treatment, Censoring at Date of Last Contact
Time Frame: From Study Initiation up to Day 672
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | LAI 590 mg QD
Number analyzed (Participants) | 206
Participants
  After Day 1 through Day 337 | 81
  After Day 1 through Day 672 | 108

16. Secondary Outcome: Number of Participants Who Received Antipseudomonal Antibiotic Treatment for Protocol Defined Pulmonary Exacerbation
Time Frame: From Study Initiation up to Day 700
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | LAI 590 mg QD
Number analyzed (Participants) | 206
Participants
  Number of patients with the event through Day 700 | 148
  Number censored | 58

ADVERSE EVENTS:
Time Frame: From enrollment up to a maximum of 672 Days (end of study, year 2)
Groups:
- LAI 590 mg QD: Liposomal amikacin for inhalation: - Liposomal amikacin for inhalation is provided as a sterile aqueous liposomal dispersion for inhalation via nebulization.
  * 590 mg of liposomal amikacin for inhalation is administered once daily using the PARI Investigational eFlow® Nebulizer.
  * Administration time is approximately 13 minutes.
  * Liposomal amikacin for inhalation will be administered in two consecutive extension periods, each consisting of 6 cycles for a total of 12 cycles. Each cycle consists of 28 days on-treatment followed by 28 days off-treatment.
Arm/Group | LAI 590 mg QD
All-Cause Mortality (participants affected / at risk) | 1/206
Serious Adverse Events (participants affected / at risk) | 92/206
Other Adverse Events (participants affected / at risk) | 167/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAI 590 mg QD (N=206)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 81 (139)
Appendicitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Lung infection pseudomonal (Infections and infestations) | 1 (1)
Measles (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 2 (2)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Cerebrospinal fluid rhinorrhoea (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Neurological symptom (Nervous system disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Pulmonary function test decreased (Investigations) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAI 590 mg QD (N=206)
Diarrhoea (Gastrointestinal disorders) | 15 (23)
Pyrexia (General disorders) | 13 (15)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 129 (359)
Nasopharyngitis (Infections and infestations) | 52 (88)
Upper respiratory tract infection (Infections and infestations) | 32 (64)
Pharyngitis (Infections and infestations) | 18 (20)
Rhinitis (Infections and infestations) | 16 (19)
Sinusitis (Infections and infestations) | 15 (18)
Viral infection (Infections and infestations) | 15 (15)
Bronchitis (Infections and infestations) | 11 (15)
Headache (Nervous system disorders) | 19 (25)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 30 (69)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (45)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 25 (40)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the signed Investigator Agreement in the protocol and protocol amendments, the PI agreed that the information presented in the study protocol is confidential, and assured that no information based on the conduct of the study was released without prior Insmed Incorporated Consent, unless the requirement is superseded by the Food and Drug Administration or other regulatory authority.